CLINICAL TRIAL: NCT04451850
Title: Heart Rate Variability (HRV) as a Marker of Treatment Response in Pulmonary Arterial Hypertension (PAH)
Brief Title: HRV as a Marker of Treatment Response in PAH Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Arun Jose, Assistant Professor of Medicine, University of Cincinnati
Other Study IDs: 2019-1371
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Noninvasive actigraphy monitor — Noninvasive chest-mounted actigraphic device to be worn for 2 hour intervals two times per week during the six month study participation.
  Other Names: Polar H10 Heart Rate Monitor

SUMMARY:
This is a prospective longitudinal cohort study to determine the value of HRV obtained using noninvasive actigraphy to quantify the response to pulmonary vasodilator therapy in newly diagnosed PAH patients

DETAILED DESCRIPTION:
This single center prospective longitudinal cohort study will take place at the University of Cincinnati (UC). We will screen adult patients newly diagnosed with PAH and placed on targeted pulmonary vasodilator therapy by their treating physician for enrollment.

We will enroll 35 eligible participants over a two-year period. HRV will be measured using the Polar™ H10 wearable chest actigraphy device in conjunction with analytic software to capture HRV data.

After enrollment and completion of the baseline visit, study participants will receive chest actigraphy device to measure their heart rate for a two hour period twice a week during study participation. Follow up research visits will be conducted at one-month, 3-months, and 6-months to sync the actigraphy device and assess any AE's.

In-between these visits, study staff will communicate with participants at two weeks, two months, 4 months, and 5 months, to identify and address any issues with study actigraphic device, assess any adverse events and maintain regular contact with study participants.

Throughout study participation, subjects will continue routine clinical care at the direction of their treating physician as needed.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (ages 18-70) of any functional class with a new diagnosis of PAH (World health Organization Group 1) placed on targeted therapy
* Eligible PAH etiologies include idiopathic PAH, associated with connective tissue disease, human immunodeficiency virus, hereditary, or portopulmonary hypertension
* Right heart catheterization (RHC) hemodynamics with a mean pulmonary arterial pressure >=20 millimetres of mercury at rest, a pulmonary capillary wedge pressure <= 15 millimetres of mercury, and a pulmonary vascular resistance >= 3 woods units

Exclusion Criteria:

* Inability to undergo (non-contrast) Magnetic Resonance Imaging (MRI) testing
* On chronotropic agents (Beta-Blockers, anti-arrhythmic medications, etc.) that could affect the calculation and interpretation of HRV measures
* Conditions that could affect the accuracy of MRI imaging, including a history previously repaired or unrepaired congenital heart defects, ventricular or atrial septal defects, or other anatomic cardiac abnormalities)
* Inability to complete a six-minute walk test
* Currently being on targeted PAH therapy at the time of consent and enrollment
* Thyroid disease, known arrhythmias in the past six months, uncontrolled anemia with a hemoglobin less than 7 grams per deciliter, untreated coronary artery disease or a diagnosis of myocardial infarction in the past 6 months, the presence of a cardiac pacemaker
* Clinically significant lung disease (including pulmonary function testing forced vital capacity < 60%), a positive ventilation/perfusion scan, uncontrolled sleep apnea not adherent with noninvasive positive pressure ventilation
* Unable to consent, pregnant women, and prisoners.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at the University of Cincinnati PAH Clinic in Cincinnati, Ohio
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HRV via RMSSD | 6 months
  Change from baseline in Root Mean Squared Successive Differences (RMSSD) measure of Heart Rate variability in patients on targeted therapy

SECONDARY OUTCOMES:
Change from baseline in HRV via SDNN | 6 months
  Change from baseline in Standard Deviation of N-to-N (SDNN) measure of Heart Rate Variability in patients on targeted therapy
Correlation with Cardiac Magnetic Resonance Imaging Variables | 6 months
  Correlation between RMSSD and SDNN with key cardiac Magnetic Resonance Imaging Variables of PAH disease, the Right Ventricular Stroke Volume
Correlation with NTproBNP | 6 months
  Correlation between RMSSD and SDNN with N-terminal Pro-B-Type Natriuretic Peptide (NTproBNP), a marker of PAH disease severity and treatment response
Correlation with REVEAL 2.0 Risk Score | 6 months
  Correlation between RMSSD and SDNN with the REVEAL 2.0 Risk score, a measure of PAH prognosis
Correlation with CAMPHOR Quality of Life Score | 6 months
  Correlation between RMSSD and SDNN with the Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) score, a 3-domain quality of life assessment tool specific to PAH patients

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jose, MD, MS, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heresi GA, Dweik RA. Strengths and limitations of the six-minute-walk test: a model biomarker study in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2011 May 1;183(9):1122-4. doi: 10.1164/rccm.201012-2079ED. No abstract available. PMID 21531951
- [Background] Ulrich S, Fischler M, Speich R, Bloch KE. Wrist actigraphy predicts outcome in patients with pulmonary hypertension. Respiration. 2013;86(1):45-51. doi: 10.1159/000342351. Epub 2012 Dec 11. PMID 23234873
- [Background] Pugh ME, Buchowski MS, Robbins IM, Newman JH, Hemnes AR. Physical activity limitation as measured by accelerometry in pulmonary arterial hypertension. Chest. 2012 Dec;142(6):1391-1398. doi: 10.1378/chest.12-0150. PMID 22576635